CLINICAL TRIAL: NCT04023175
Title: In Office Versus Telemedicine Preoperative Visit: a Randomized Controlled Trial
Brief Title: In Office Versus Telemedicine Preoperative Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 05-19-30E
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2021-06

CONDITIONS: Telemedicine
Keywords: Virtual visit; Preoperative counseling; Preoperative preparedness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In office (Active Comparator): Patients will undergo our standard in office preoperative counseling.
  Interventions: Other: In office preoperative counseling
- Virtual visit (Experimental): Patients will undergo preoperative counseling using telemedicine virtual visits.
  Interventions: Other: Telemedicine preoperative counseling

INTERVENTIONS:
Other: Telemedicine preoperative counseling — The telemedicine visit will be completed using an Atrium Health approved virtual visit platform.
  Arms: Virtual visit
Other: In office preoperative counseling — This includes our standard preoperative counseling located at the Women's Center for Pelvic Health
  Arms: In office

SUMMARY:
This is a randomized controlled trial evaluating in office versus telemedicine preoperative counseling visits based on patient preparedness for surgery and patient satisfaction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE To determine whether preoperative telemedicine appointments are non-inferior to in-office visits based on patient preoperative preparedness in women undergoing pelvic surgery as measured by a preoperative preparedness survey.

SECONDARY OBJECTIVES

1. Evaluate patient satisfaction using the S-CAHPS survey
2. Calculate the duration of visit for patient (minutes)
3. Calculate the duration of visit for provider (minutes)
4. Estimate round trip travel distance from patient home to clinic (miles)
5. Evaluate the number of office contacts from date of preoperative counseling to 6 weeks postoperatively.

   1. Patient initiated calls
   2. Nurse initiated calls
   3. Scheduled office visits
   4. Add on office visits
6. Evaluate canceled, no-show, and late visits
7. Calculate value proposition metrics for Atrium Health System

PREOPERATIVE PERIOD All consecutive patients planning to undergo pelvic surgery who require a preoperative visit will be identified, screened, and approached for participation in the study. Participants who do not meet the inclusion and exclusion criteria will be considered screen failures. Screen failures will be captured and the cause for screen failure will be documented.

Verbal consent will be obtained and accurate email address will be confirmed. Eligible subjects will be randomized using a computer-generated randomization scheme with patients assigned in a 1:1 ratio to either:

Study Group: Telemedicine preoperative counseling with a Female Pelvic Medicine and Reconstructive Surgery (FPMRS) fellow

Control Group: Standard in-office preoperative counseling with a FPMRS fellow

The allocation sequence will be in numerical, sealed, opaque envelopes. An envelope will be retrieved at the time of consent. The surgical scheduler will then schedule the patient for their allocated preoperative visit.

Prior to their preoperative visit, participants in both groups will be emailed copies of the office Enhanced Recovery After Surgery informational booklet and International Urogynecology Association (IUGA) patient information handouts pertinent to their surgery. The preoperative visit at Women's Center for Pelvic Health (WCPH) is a counseling visit to review informed consent. Preoperative medical evaluation is accomplished through the Carolinas Hospitalist Group preoperative clinic or with the patient's primary care provider. Patients who require preoperative medical clearance will be scheduled for a preoperative visit with the Carolinas Hospitalist Group or their primary care provider in addition to their preoperative visit with the WCPH. These visits will be documented in the total office visit data collection.

Women in the Telemedicine group will check in for their preoperative visit via an Atrium Information Systems (IS) approved virtual communication platform at the scheduled date and time. They will undergo preoperative counseling following a standardized checklist format. After telemedicine counseling has concluded, participants will be emailed a REDCap survey link to complete a survey regarding their preparation for surgery. If a participant has not completed the survey by the next business day, an email reminder will be sent to their email address on file. If they have not completed the survey within 2 business days, they will be contacted by phone for reminder. If a participant in the Telemedicine group ultimately elects to have an in-office preoperative visit, they will be scheduled for in-office visit and analyzed as intention-to-treat.

Women in the In-office group will present to WCPH for preoperative in-person counseling following a standardized checklist format. After in-office counseling has concluded, participants will be asked to complete a survey regarding preparation for surgery via a REDCap survey link on an Atrium IS approved iPad prior to leaving the office.

PERIOPERATIVE PERIOD Participants will present to Mercy Hospital or One Day Surgery Center for their scheduled surgery. All participants will receive routine care according to the gynecologic enhanced recovery perioperative protocol. The gynecologic enhanced recovery perioperative protocol is a multimodal perioperative care pathway designed to achieve early recovery after surgery by maintaining preoperative organ function and reducing the physical stress of surgery on the body. This protocol includes many components including allowing patients to drink clear liquids up to 2 hours prior to their surgery, maintaining euvolemia intraoperatively, and early return to normal diet and activity after surgery. All patients undergoing pelvic reconstructive surgery are scheduled for the enhanced recovery protocol, except for women having only minor procedures such as mid-urethral sling placement or cystoscopy.

POSTOPERATIVE PERIOD All participants will undergo routine postoperative care. They will be scheduled for an in-office postoperative visit, on average 1-2 weeks after surgery and then again at 6 weeks after surgery per our office standard practice. Following their 2-week postoperative visit, women will be asked to complete the preoperative subsection of the Surgical-CAHPS survey to evaluate patient satisfaction. This will be given to all patients prior to leaving the office. If a patient does not present to their 2-week postoperative appointment, they will be mailed a paper copy of the preoperative subsection of the S-CAHPS and asked to return this via prepaid postage.

Following the 6 week postoperative visit, secondary data will then be extracted from the electronic medical record (EMR) via manual chart view.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18 and greater
* Visit location in North Carolina
* Planning to undergo pelvic surgery at Mercy Hospital or One Day Surgery Center
* Scheduled for enhanced recovery perioperative protocol
* Require a preoperative visit
* Access to internet and a virtual visit capable device
* Telephone access

Exclusion Criteria:

* Non-English speaking
* Inability to provide consent/decisionally impaired
* Auditory impairment
* Required preoperative in-office procedure such as endometrial biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-07-27 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Braxton, MD, Principal Investigator — Novant Health
Locations (1):
- Women's Center for Pelvic Health-Mercy, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seidel JE, Beck CA, Pocobelli G, Lemaire JB, Bugar JM, Quan H, Ghali WA. Location of residence associated with the likelihood of patient visit to the preoperative assessment clinic. BMC Health Serv Res. 2006 Feb 22;6:13. doi: 10.1186/1472-6963-6-13. PMID 16504058
- [Background] 2. Health Resources and Services Administration. (https://www.hrsa.gov/rural-health/telehealth/index.html) May 2019.
- [Background] LaMonte MP, Bahouth MN, Hu P, Pathan MY, Yarbrough KL, Gunawardane R, Crarey P, Page W. Telemedicine for acute stroke: triumphs and pitfalls. Stroke. 2003 Mar;34(3):725-8. doi: 10.1161/01.STR.0000056945.36583.37. Epub 2003 Jan 30. PMID 12624298
- [Background] Platts-Mills TF, Hendey GW, Ferguson B. Teleradiology interpretations of emergency department computed tomography scans. J Emerg Med. 2010 Feb;38(2):188-95. doi: 10.1016/j.jemermed.2008.01.015. Epub 2008 Sep 23. PMID 18814996
- [Background] Asiri A, AlBishi S, AlMadani W, ElMetwally A, Househ M. The Use of Telemedicine in Surgical Care: a Systematic Review. Acta Inform Med. 2018 Oct;26(3):201-206. doi: 10.5455/aim.2018.26.201-206. PMID 30515013
- [Background] Applegate RL 2nd, Gildea B, Patchin R, Rook JL, Wolford B, Nyirady J, Dawes TA, Faltys J, Ramsingh DS, Stier G. Telemedicine pre-anesthesia evaluation: a randomized pilot trial. Telemed J E Health. 2013 Mar;19(3):211-6. doi: 10.1089/tmj.2012.0132. Epub 2013 Feb 5. PMID 23384334
- [Background] Lozada MJ, Nguyen JT, Abouleish A, Prough D, Przkora R. Patient preference for the pre-anesthesia evaluation: Telephone versus in-office assessment. J Clin Anesth. 2016 Jun;31:145-8. doi: 10.1016/j.jclinane.2015.12.040. Epub 2016 Apr 15. PMID 27185698
- [Background] Nikolian VC, Williams AM, Jacobs BN, Kemp MT, Wilson JK, Mulholland MW, Alam HB. Pilot Study to Evaluate the Safety, Feasibility, and Financial Implications of a Postoperative Telemedicine Program. Ann Surg. 2018 Oct;268(4):700-707. doi: 10.1097/SLA.0000000000002931. PMID 30095477
- [Background] Soegaard Ballester JM, Scott MF, Owei L, Neylan C, Hanson CW, Morris JB. Patient preference for time-saving telehealth postoperative visits after routine surgery in an urban setting. Surgery. 2018 Apr;163(4):672-679. doi: 10.1016/j.surg.2017.08.015. Epub 2018 Feb 3. PMID 29398042
- [Background] Myers EM, Rustowicz L, Wells D, Kidd JB, Jannelli ML, Connolly A, Wu JM. Internet Use Among Urogynecology Patients in North Carolina. Female Pelvic Med Reconstr Surg. 2015 Sep-Oct;21(5):269-72. doi: 10.1097/SPV.0000000000000163. PMID 25730431
- [Background] Mazloomdoost D, Kanter G, Chan RC, Deveaneau N, Wyman AM, Von Bargen EC, Chaudhry Z, Elshatanoufy S, Miranne JM, Chu CM, Pauls RN, Arya LA, Antosh DD. Social networking and Internet use among pelvic floor patients: a multicenter survey. Am J Obstet Gynecol. 2016 Nov;215(5):654.e1-654.e10. doi: 10.1016/j.ajog.2016.06.011. Epub 2016 Jun 16. PMID 27319368
- [Background] Thompson, J MD et al. Outpatient visits versus telephone interviews for postoperative care: A randomized controlled trial (OPTIONS). [abstract] In: Proceedings of the 39th Annual Scientific Meeting of the American Urogynecologic Society; 2018 Oct 9-13; Chicago, IL Paper nr 1
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686

RESULTS

PARTICIPANT FLOW:
Groups:
- In Office: Patients underwent standard in office preoperative counseling.
  In office preoperative counseling: This includes our standard preoperative counseling located at the Women's Center for Pelvic Health
- Virtual Visit: Patients underwent preoperative counseling using telehealth virtual visits.
  Telemedicine preoperative counseling: The telemedicine visit was completed using an Atrium Health approved virtual visit platform.
Period: Overall Study
Arm/Group | In Office | Virtual Visit
Started | 59 | 59
Completed | 53 | 48
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In Office | Virtual Visit | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.5) | 59.0 (10.9) | 60.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 58 | 58 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 52 | 50 | 102
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Preoperative Preparedness
Description: To determine whether preoperative telemedicine appointments are non-inferior to in-office visits based on patient preoperative preparedness in women undergoing pelvic surgery as measured by a preoperative preparedness survey.
  Preoperative Preparedness Questionnaire ranges from 11 to 66 points with higher scores equaling greater patient preparedness.
Time Frame: 1-7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
units on a scale | 63.0 (3.6) | 62.5 (4.6)

2. Secondary Outcome: Patient Satisfaction
Description: Patients will complete the preoperative portion of the Consumer Assessment of Healthcare Providers and Systems Surgical Care Survey (S-CAHPS) at the 2-week postoperative visit. S-CAHPS is a validated standardized questionnaire for adults developed by the American College of Surgeons (ACS). There are various ways to score. We elected to measure total composite scores of the perioperative SCAHPS subsection ranging from 12 to 36, with greater scores equating to higher patient satisfaction. The minimum value is 0 and maximum is 33.
Time Frame: 2 week postoperative visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
score on a scale | 30.5 (2.1) | 31.3 (1.5)

3. Secondary Outcome: Duration of Visit
Description: Each visit will be timed to evaluate patient and provider visit duration. Timing will begin for the Telemedicine group upon connection to the virtual waiting room and will conclude after all counseling is completed and the virtual visit is disconnected. The duration of virtual visit counseling time with the provider will also be calculated. Timing for the in-office group will begin at time of patient check-in at the front desk and will conclude with patient check-out.
Time Frame: at preoperative visit (1-30 days prior to surgery)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
minutes | 55.9 (18.9) | 39.3 (14.0)

4. Secondary Outcome: Round Trip Travel Distance
Description: Round trip travel distance from patient's home address to office will be evaluated via a HIPPA compliant map-based search engine for each participant.
Time Frame: at preoperative visit (1-30 days prior to surgery)
Measure: Median (Inter-Quartile Range); unit: miles
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
miles | 28 [20.0 to 46.0] | 0 [0 to 0]

5. Secondary Outcome: Office Contacts, Total Scheduled In-person Visits
Description: The total number of scheduled in-person visits in the perioperative time period including preoperative and postoperative visits..
Time Frame: perioperative time period, up to approximately 10 weeks
Measure: Median (Inter-Quartile Range); unit: visits
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
visits | 3.0 [2.00 to 3.00] | 2.0 [2.00 to 2.00]

6. Secondary Outcome: Postoperative Add on In-person Visits.
Description: Clinical visits added in the six week postoperative time period.
Time Frame: 6 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: number of visits
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
number of visits | 0 [0.0 to 1.0] | 0 [0.0 to 1.0]

7. Secondary Outcome: Postoperative Patient Initiated Phone Calls.
Description: Number of patient initiated postoperative telephone calls to the office in the six week postoperative time period.
Time Frame: 6 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: phone calls
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
phone calls | 1 [0.0 to 2.0] | 1 [1.0 to 3.0]

8. Secondary Outcome: Travel Time
Description: Patient round-trip travel time in minutes from home to preoperative visits.
Time Frame: 1 day of a preoperative visit.
Population: patient
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | In Office | Virtual Visit
Number analyzed (Participants) | 59 | 59
minutes | 66.0 [50.0 to 80.0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 6 weeks postoperatively
Arm/Group | In Office | Virtual Visit
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 9/59 | 6/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Office (N=59) | Virtual Visit (N=59)
Urinary Tract Infection (Renal and urinary disorders) | 8 (8) | 5 (5)
Intraoperative cystotomy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04023175/Prot_SAP_000.pdf